CLINICAL TRIAL: NCT01268176
Title: Meal Effects on the 25OHD3 Response to Supplemental Vitamin D3
Brief Title: The Effect of a Meal on Vitamin D Absorption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Bess Dawson-Hughes, Director, Bone Metabolism Laboratory, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2660
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; vitamin D deficiency; vitamin D absorption
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low fat meal (Active Comparator): Those subjects who receive a low fat meal prior to vitamin D3 administration
  Interventions: Dietary Supplement: cholecalciferol
- High fat meal (Active Comparator): Those subjects who receive a high fat meal prior to vitamin D3 administration
  Interventions: Dietary Supplement: cholecalciferol
- No meal (Active Comparator): Those subjects who do not receive a meal and continue to fast. They only receive the vitamin D3 dose.
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 50,000 IU once per month for 3 months
  Other Names: vitamin D3

SUMMARY:
This study seeks to determine if vitamin D3 absorption in healthy adults will be enhanced in the presence of a meal and if the enhancement will be greater when the meal is low as opposed to high in fat content. The enhancement will result from increased vitamin D absorption. The investigators will test this hypothesis by pursuing the following aims in a 3-mo trial in which up to 70 healthy men and women will be randomized to one of the following meal conditions under which they will take a monthly oral dose of 50,000 IU of vitamin D3: no meal (fasting), a low fat meal, or a high fat meal. The Primary Aim is to identify the meal condition (fasting, low-fat, or high-fat meal) under which the 25OHD3 response to supplemental vitamin D3 is greatest and most consistent. The Secondary Aim is to determine whether vitamin D3 absorption is affected by the meal condition and to determine whether the absorption of vitamin D3 predicts the longer-term 25OHD3 response to supplementation.

DETAILED DESCRIPTION:
Vitamin D supplements are increasingly recommended to curb widespread deficiency. Decreasing the variability in 25OHD responses to supplemental vitamin D would make the supplementation process more predictable, and thereby reduce the number of 25OHD measurements and dose adjustments that are needed to achieve the targeted 25OHD level. This study seeks to identify potential sources of variability in the 25OHD3 response to supplemental vitamin D3 that are plausible based on rat studies, but have not been explored in humans. The investigators hypothesize that the serum 25OHD3 response to supplemental vitamin D3 in healthy adults will be enhanced in the presence of a meal and the enhancement will be greater when the meal is low as opposed to high in fat content. The enhancement will result from increased vitamin D absorption. The investigators will test this hypothesis by pursuing the following aims in a 3-mo trial in which up to 70 healthy men and women will be randomized to one of the following meal conditions under which they will take a monthly oral dose of 50,000 IU of vitamin D3: no meal (fasting), a low fat meal, or an iso-caloric high fat meal. Serum 25OHD3 will be measured at baseline and after 1 and 3 mo. A serum vitamin D3 absorption test will be performed in each subject after the first dose of vitamin D. The Primary Aim is to identify the meal condition (fasting, low-fat, or high-fat meal) under which the 25OHD3 response to supplemental vitamin D3 is greatest and most consistent. The Secondary Aim is to determine whether vitamin D3 absorption is affected by the meal condition and to determine whether the absorption of vitamin D3 predicts the longer-term 25OHD3 response to supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50 to 69
* BMI ≥ 18.5 and ≤ 27.9 kg/m2
* those taking ≤ 400 IU/day of vitamin D3 and ≤ 1000 mg calcium/day
* those who participate must agree not to change their dietary or supplemental vitamin D or calcium intake during the study
* no use of tanning salons
* no travel south of latitude 34 degrees north during the study

Exclusion Criteria:

General:

1. A screening 25OHD level ≤8 or ≥ 25 ng/ml
2. An abnormal serum calcium (reference range is 8.3 -10.2 mg/dl)
3. A screening spot urinary calcium:creatinine ratio > 0.325
4. Greater than 2 drinks of alcohol a day.
5. BMI <18.5 and >27.9 kg/m2
6. Menses within the last year (women)
7. Age <50 and > 69 years
8. Allergy to egg
9. A blood donation in the last 2 months (increases likelihood of anemia)
10. Non-English speaking subjects will not be enrolled.
11. Other abnormalities in screening labs, at the discretion of the study physician (PI)

Medications:

1. Subjects must agree not to take more than 400 IU per day of vitamin D as supplement or cod liver oil during the study
2. Topical vitamin D preparations
3. Oral estrogen or estrogen patch use in the last 6 months
4. Regular antacid use (>2 times per week)
5. Sucralfate
6. Acarbose/miglitol
7. PPIs - prescription: lansoprazole (Prevacid), omeprazole (Prilosec and Zegerid), esomeprazole (Nexium), rabeprazole (Aciphex), pantoprazole (Protonix); over-the-counter: lansoprazole (Prevacid 24), omeprazole (Prilosec OTC), zegerid OTC (Equate), omeprazole magnesium
8. H2 blockers - prescription: cimetidine (Tagamet), famotidine (Pepsid), nizatidine (Axid), rantidine hydrochloride (Zantac), dexlansoprazole (Kapidex); over the counter: cimetidine (Tagamet-HB, Equate), famotidine (Pepcid-AC, Pepcid Complete), rantidine hydrochloride (Zantac, Wal-Zan, Equate)
9. Drugs that alter fat and cholesterol handling - xenical and alli (Orlistat), cholestyramine (Questran, LoCholest, Prevalite), Zetia
10. Drugs that alter 25OHD metabolism - Antiseizure drugs phenobarbitol and phenytoin (Dilantin), oral glucocorticoids
11. Calcium supplement use >1000 mg/day

Diseases:

1. Active parathyroid disease
2. Sarcoidosis
3. Peptic ulcers or esophageal stricture
4. Active malignancy (other than basal cell cancer of the skin) or cancer therapy in the last year
5. Advanced kidney disease (creatinine clearance <30 ml/min calculated from serum creatinine with use of the Modification of Diet in Renal Disease (MDRD) Study equation
6. Kidney stones in the last 5 years.
7. Liver disease
8. Zollinger-Ellison syndrome
9. Known achlorhydria or small bowel overgrowth
10. Malabsorption
11. Diseases associated with fat malabsorption - liver disease, cystic fibrosis, Celiac disease, bariatric surgery, Scleroderma, Crohn's, prior surgery involving the stomach or small bowel (appendectomy okay), gall stones or prior gall bladder surgery, pancreatitis

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
25OHD3 response to supplemental vitamin D3 | 3 months
  To identify the meal condition (fasting, low-fat, or high-fat meal) under which the 25OHD3 response to supplemental vitamin D3 is greatest and most consistent, specifically, to describe and compare changes in serum 25OHD3 concentration across the 3 groups.

SECONDARY OUTCOMES:
Change in parent vitamin D3 levels | 12 hours
  To determine whether vitamin D3 absorption is affected by the meal condition, specifically,a) to describe and compare the change in parent vitamin D3 levels over the 12-hr period following the first dose of vitamin D3 across the 3 groups and b) to determine whether the absorption of vitamin D3 at 12 hours predicts the longer-term 25OHD3 response to supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, M.D., Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Fu L, Yun F, Oczak M, Wong BY, Vieth R, Cole DE. Common genetic variants of the vitamin D binding protein (DBP) predict differences in response of serum 25-hydroxyvitamin D [25(OH)D] to vitamin D supplementation. Clin Biochem. 2009 Jul;42(10-11):1174-7. doi: 10.1016/j.clinbiochem.2009.03.008. Epub 2009 Mar 18. PMID 19302999
- [Background] Dawson-Hughes B, Harris SS, Dallal GE. Plasma calcidiol, season, and serum parathyroid hormone concentrations in healthy elderly men and women. Am J Clin Nutr. 1997 Jan;65(1):67-71. doi: 10.1093/ajcn/65.1.67. PMID 8988915
- [Background] Heaney RP, Davies KM, Chen TC, Holick MF, Barger-Lux MJ. Human serum 25-hydroxycholecalciferol response to extended oral dosing with cholecalciferol. Am J Clin Nutr. 2003 Jan;77(1):204-10. doi: 10.1093/ajcn/77.1.204. PMID 12499343
- [Background] Dawson-Hughes B, Heaney RP, Holick MF, Lips P, Meunier PJ, Vieth R. Estimates of optimal vitamin D status. Osteoporos Int. 2005 Jul;16(7):713-6. doi: 10.1007/s00198-005-1867-7. Epub 2005 Mar 18. PMID 15776217
- [Background] Hollander D, Muralidhara KS, Zimmerman A. Vitamin D-3 intestinal absorption in vivo: influence of fatty acids, bile salts, and perfusate pH on absorption. Gut. 1978 Apr;19(4):267-72. doi: 10.1136/gut.19.4.267. PMID 25826
- [Background] Mulligan GB, Licata A. Taking vitamin D with the largest meal improves absorption and results in higher serum levels of 25-hydroxyvitamin D. J Bone Miner Res. 2010 Apr;25(4):928-30. doi: 10.1002/jbmr.67. PMID 20200983
- [Background] Krall EA, Sahyoun N, Tannenbaum S, Dallal GE, Dawson-Hughes B. Effect of vitamin D intake on seasonal variations in parathyroid hormone secretion in postmenopausal women. N Engl J Med. 1989 Dec 28;321(26):1777-83. doi: 10.1056/NEJM198912283212602. PMID 2594036
- [Background] Rockell JE, Skeaff CM, Williams SM, Green TJ. Association between quantitative measures of skin color and plasma 25-hydroxyvitamin D. Osteoporos Int. 2008 Nov;19(11):1639-42. doi: 10.1007/s00198-008-0620-4. Epub 2008 Apr 12. PMID 18408879
- [Background] Vieth R, Chan PC, MacFarlane GD. Efficacy and safety of vitamin D3 intake exceeding the lowest observed adverse effect level. Am J Clin Nutr. 2001 Feb;73(2):288-94. doi: 10.1093/ajcn/73.2.288. PMID 11157326